CLINICAL TRIAL: NCT01324765
Title: Women Overcoming and Managing Adversity Now (WOMAN) Study
Acronym: WOMAN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Julian D. Ford, University of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09009-2; 2009-DD-BX-0003 (Other Grant/Funding Number: Department of Justice)
Record Dates: First submitted 2010-09-23; First posted 2011-03-29 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Posttraumatic Stress Disorder; PTSD
Keywords: Women; PTSD; Group Therapy; Incarceration
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TARGET (Experimental): 12-session affect regulation therapy for PTSD
  Interventions: Behavioral: TARGET
- SGT (Active Comparator): 12 session supportive group therapy
  Interventions: Behavioral: SGT

INTERVENTIONS:
Behavioral: TARGET — 12-session group therapy twice weekly 6 weeks
  Arms: TARGET
Behavioral: SGT — 12 sessions supportive group therapy twice weekly 6 weeks
  Arms: SGT

SUMMARY:
The goal of the study is to evaluate the efficacy of a two therapeutic models designed to enhance women's skills for managing reactive emotions in their current lives as well as to educate them about how using these skills can enhance their personal effectiveness and help them to gain control of post-traumatic stress reactions. The interventions adaptations of a manualized psychotherapy that has shown promise with adults with complex Posttraumatic Stress Disorder (PTSD) (Trauma Affect Regulation: Guide for Education and Therapy; TARGET) compared to a supportive group therapy (SGT) that has been found to have modest benefits with women survivors of childhood abuse (Wallis, 2002).

DETAILED DESCRIPTION:
In a randomized treatment design, we will compare offenders receiving skills-based intervention (TARGET) and those receiving a similar amount of supportive intervention (SGT). We will assess the efficacy of treatment by determining if those receiving the TARGET skills training show an improvement in functionality, as compared to those receiving only supportive intervention. We will measure this by analyzing PTSD symptoms, psychological distress, psychosocial functioning, and social/legal adjustment and services using structured interviews, self-report questionnaires and qualitative questions. Questionnaires are listed below in the outcome measure's section. We will collect follow-up data on program participants who successfully finish the program at York. For those offenders who discharge into the community directly from York, we will collect follow-up data on program participants through CDOC Parole or Probation records. Statistically we anticipate a medium effect size difference between the treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated, release not expected within 6 months
* Probable PTSD on PC-PTSD screen and PTSD by CAPS interview

Exclusion Criteria

* Clinically significant psychopathy (PCL-SV severe range)
* Unable to comprehend study materials (Mini-Mental Status Exam Orientation, Attention, and Recall sections total score <15).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
PTSD | Post-therapy (within 2 weeks)
  PTSD symptom severity, Clinician Administered PTSD Scale
PTSD | 3-4 Month Post-therapy Follow-up
  PTSD symptom severity, Clinician Administered PTSD Scale

SECONDARY OUTCOMES:
Emotion Regulation | Post-therapy (within 2 weeks)
  Negative Mood Regulation Scale
Trauma-related symptoms | Post-therapy (within 2 weeks)
  Trauma Symptom Inventory (TSI; Briere, 1995). The TSI is a reliable and validated 100-item measure that generates composite scores for trauma (PTSD symptoms), self (self-regulation problems), and dysphoria (depression, anxiety, anger symptoms).
Mental health symptoms, well-being, and self-harm | Post-therapy (within 2 weeks)
  CORE-OM is a 34-item self-report measure reliably and validly assessing current psychiatric symptom severity, risk of harm to self or others, social functioning, and subjective well being
Emotion Regulation | 3-4 Month Post-therapy Follow-up
  Negative Mood Regulation Scale
Trauma-related Symptoms | 3-4 Month Post-therapy Follow-up
  Trauma Symptom Inventory
Mental health symptoms, well-being, and self-harm | 3-4 Month Post-therapy Follow-up
  CORE-OM 34-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Julian D Ford, Ph.D., Principal Investigator — UConn Health
Locations (1):
- York Correctional Institution, Niantic, Connecticut, United States